CLINICAL TRIAL: NCT01973556
Title: Pharmacist-Physician Collaborative Medication Therapy Management Services (MTMS) Demonstration Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jan Hirsch, Associate Professor Clinical Pharmacy, University of California, San Diego
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20095191; 100492 (Other: UCSD Human Subjects Protection Program)
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacist-Physician Collaborative Medication Management (Experimental): Pharmacist-Physician Collaborative Medication Management
  Interventions: Other: Pharmacist-Physician Collaborative Medication Therapy Management
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Pharmacist-Physician Collaborative Medication Therapy Management
  Arms: Pharmacist-Physician Collaborative Medication Management

SUMMARY:
Patients managed by a newly formed pharmacist-physician medication therapy management team in a university primary care clinic will have better blood pressure control than patients receiving usual care.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or over
* diagnosis of hypertension with most recent blood pressure >140/90 mmHg or blood pressure >130/80 mmHg if patients also had diabetes mellitus
* treated with at least one anti-hypertensive medication
* continuous active patient (at least one visit) of the clinic for at least the past 6 months (1/1/2010-6/31/2010)
* English speaking
* Able to complete questionnaires in English.

Exclusion Criteria:

-do not meet provisions of the clinical collaborative agreement protocol in the judgment of the patient's physician or the clinical pharmacist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Hirsch JD, Steers N, Adler DS, Kuo GM, Morello CM, Lang M, Singh RF, Wood Y, Kaplan RM, Mangione CM. Primary care-based, pharmacist-physician collaborative medication-therapy management of hypertension: a randomized, pragmatic trial. Clin Ther. 2014 Sep 1;36(9):1244-54. doi: 10.1016/j.clinthera.2014.06.030. Epub 2014 Jul 30. PMID 25085406